CLINICAL TRIAL: NCT06780514
Title: Cardiopulmonary Exercise Testing in Girls (8-18y) with Turner Sydrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2023-0632
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Turner Syndrome
Keywords: Cardiopulmonary exercise test
MeSH Terms: conditions — Turner Syndrome | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test — To our knowledge, this is the first study to perform CPET's in Turner Girls aged <18 years
  Other Names: CPET; cyclo-ergometry

SUMMARY:
The goal of this clinical trial is to have a beter insight in the exercise tolerance in girls with Turner Syndrome aged 8-18 years . The main question it aims to answer is:

Is there a difference in VO2 max comparing Turner syndrome girls with standard values? How do cardiovascular parameters change during exercise (heart rate, bloodpressure, ...)

Participants will perform a cyclo-ergometry in a standardised way.

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome girls aged 8-18 years old

Exclusion Criteria:

* Severe mental impairement making it impossible to perform an exercise test

Ages: 8 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
VO2 max | Whitin a week after the CPET
  VO2 max is the maximum volume (V) of oxygen (O2) your body can process during exercise

SECONDARY OUTCOMES:
Bloodpressure | Whitin a week after the CPET
Heart rate | Whitin a week after the CPET

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No